CLINICAL TRIAL: NCT02611739
Title: Using a Humanoid Robot to Reduce Procedural Pain and Distress in Children With Cancer: A Pilot Randomized Controlled Trial
Brief Title: Medi-Port Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, Clinical Nurse Specialist/NP, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000049494
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Actively Undergoing Cancer Treatment; 4-9 Years of Age; At Least 1 Month From Diagnosis; Able to Speak and Understand English; Presenting to Clinic for at Least a 2nd Subcutaneous Port Needle Insertion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Children in the experimental treatment condition will sit in front of the nurse and beside (or on the lap) of a parent. Medi-Port (humanoid robot) will be positioned beside the child (at eye-level) and will execute a pre-programmed series of behaviours to distract the child before, during, and after the SCP needle insertion. The nurse will insert the needle according to hospital procedures, using minimal distraction (e.g., "What's on TV?"). The estimated time for port procedures and completion of the needle insertion will range from 10-30 minutes. The total estimated time which includes the completion of surveys and questionnaires on the pain intensity of the SCP needle insertion procedure and acceptability of Medi-port will be approximately 1 hour. There will be no follow-up visits.
  Interventions: Device: Medi-Port
- Control Group (Active Comparator): Following consent and randomization, children in the (control) usual care condition will sit in front of the nurse and beside (or on the lap) of a parent. Medi-Port (humanoid robot) will be positioned beside the child (at eye-level) and will execute a standard set of dancing movements only. The nurse will insert the needle according to hospital procedures, using minimal distraction (e.g., "What's on TV?"). The estimated time for port procedures and completion of the needle insertion will range from 10-30 minutes. The total estimated time which includes the completion of surveys and questionnaires on the pain intensity of the SCP needle insertion procedure and acceptability of Medi-port will be approximately 1 hour. There will be no follow-up visits.
  Interventions: Device: Medi-Port

INTERVENTIONS:
Device: Medi-Port — Treatment
  Arms: Intervention Group
Device: Medi-Port — Control
  Arms: Control Group

SUMMARY:
Pain is a frequent and significant problem related to cancer-directed treatment in children. Children with cancer often cite needle procedures as the most distressing experience caused by cancer and its treatment. Recently it has been shown that an interactive humanoid robot is capable of facilitating distraction and reducing distress during childhood immunizations. Our research objectives are to: (1) assess the feasibility of implementing the robot (Medi-Port) for effectiveness testing in a future RCT (measured as implementation outcomes) and (2) determine treatment effectiveness estimates (measured as preliminary effectiveness outcomes), compared to standard medical care.

DETAILED DESCRIPTION:
A sample of 40 children with cancer between the ages of 4-9 years (20 participants per treatment arm; 10 boys and 10 girls per treatment arm) will be recruited. The feasibility of the trial protocol to evaluate the impact of distraction via the humanoid robot on pain intensity and distress during SCP needle insertion compared to an active control in children with cancer will be explored. The effectiveness outcome includes the examination of the robot programmed to distract children during the procedure, reduce pain intensity and distress compared to an active control intervention (i.e. dancing robot).

ELIGIBILITY:
Inclusion Criteria:

* 4-9 years
* able to speak and understand English,
* actively undergoing cancer treatment
* presenting to clinic for at least a 2nd subcutaneous port needle insertion
* being at least 1 month from diagnosis.

Exclusion Criteria:

* visual, auditory or cognitive impairments precluding interaction with Medi-Port
* end-of-life patients
* patients who are nil per os pre-sedation.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Accrual rates | 12 months
  Accrual rates will be captured by recording data related to the number of eligible children per recruitment day, reasons for ineligibility, and reasons for non-participation.
Acceptability | 12 months
  Acceptability will be measured using the Medi-Port Satisfaction Questionnaire completed by children, parent, and nurses that will collect data on acceptability, perceived utility of pain reducing procedures, and recommendations for changes related to the needle insertion experience.
Outcome measure feasibility | 12 months
  Outcome measure feasibility will be measured as the percentage of completed outcome measures at baseline and study completion (100% when all questionnaires are completed) and will be recorded on Medi-Port Activity Log.
Technical difficulties | 12 months
  Technical difficulties (occurrence and description) will be captured using the Medi-Port Intervention Log, designed to record data.
Practical difficulties | 12 months
  Practical difficulties will be captured using the Medi-Port Intervention Log, designed to record data.
Time | 12 months
  Practical difficulties will be captured using the Medi-Port Intervention Log, designed to record data.

SECONDARY OUTCOMES:
Pain intensity | 12 months
  Pain intensity (both retrospectively for previous SCP access and after the study procedures) will be measured. Children will self-report their pain and parents, nurses, and the researcher will use proxy-reporting in rating children's pain. Children will use the Faces Pain Scale-Revised (FPS-R) which has been validated in children 4 years and older. Parents, nurses, and the researcher will use an 11-point numerical rating scale (NRS), with verbal anchors of "no pain at all" at 0 and "the most pain you can imagine this child having" at 10.
Distress | 12 months
  Distress (both retrospectively for previous SCP access and after the study procedures will be measured). Children will retrospectively report fear using the Children's Fear Scale (CFS), which is a visual scale with established psychometrics in children 5-10 years. Parents will retrospectively report pain using an 11-point NRS. Distress during the study SCP access will be measured using the observer-rated Behavioral Approach-Avoidance Scale (BAADS). The same 2 trained research team members will code video-recordings from all SCP needle insertions using the BAADS. Child distress behaviours will be scored at specific steps during the procedure: 1) nurse movement towards the child 2) pre-procedure skin sterilization 3) SCP position assessment by nurse 4) needle insertion 5) sterile dressing application.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stinson, RN, PhD, Principal Investigator — The Hospital for Sick Children; Paul Nathan, MD, Principal Investigator — The Hospital for Sick Children; Tanya Beran, PhD, RPsych, Principal Investigator — University of Calgary; Lindsay Jibb, RN, MSc, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jibb LA, Birnie KA, Nathan PC, Beran TN, Hum V, Victor JC, Stinson JN. Using the MEDiPORT humanoid robot to reduce procedural pain and distress in children with cancer: A pilot randomized controlled trial. Pediatr Blood Cancer. 2018 Sep;65(9):e27242. doi: 10.1002/pbc.27242. Epub 2018 Jun 12. PMID 29893482